CLINICAL TRIAL: NCT06327529
Title: Zinc and Iron Absorption From Common Beans in Young Adult Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2101814
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Zinc Absorption; Iron Absorption
Keywords: zinc; iron; absorption; phytate; polyphenols; beans
MeSH Terms: interventions — atrial natriuretic factor (4-23)NH2, de-Gln(18)-de-Ser(19)-de-Gly(20,22)-de-Leu(21)-

STUDY DESIGN:
Intervention Model Description: A four arm multi-tracer non-randomized crossover design
Who Masked: Participant
Masking Description: Study participants will be masked to the type of bean that they will be receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bean Variety 1 (Experimental): Enriched with Zinc-67, Iron-57
  Interventions: Other: SER 118
- Bean Variety 2 (Experimental): Enriched with Zinc-70, Iron-58
  Interventions: Other: LMP 1001
- Bean Variety 3 (Experimental): Enriched with Zinc-67, Iron-57
  Interventions: Other: LPA 586
- Bean Variety 4 (Experimental): Enriched with Zinc-70, Iron-58
  Interventions: Other: KAT B1

INTERVENTIONS:
Other: SER 118 — Bean High in Phytic Acid and High in Inhibitory Polyphenols
  Arms: Bean Variety 1
Other: LMP 1001 — Bean Low in Phytic Acid and High in Inhibitory Polyphenols
  Arms: Bean Variety 2
Other: LPA 586 — Bean Low in Phytic Acid and Low in Inhibitory Polyphenols
  Arms: Bean Variety 3
Other: KAT B1 — Bean High in Phytic Acid and Low in Inhibitory Polyphenols
  Arms: Bean Variety 4

SUMMARY:
Fifteen female study participants will be enrolled in a randomized crossover study to measure fractional and total zinc and iron absorption from four common bean (Phaseolus vulgaris) varieties with varying phytate and polyphenolic contents. Phytate, the storage form of phosphorus in plants, and polyphenols, which contribute to the varied colors of common beans, are natural components of the beans and can reduce zinc and iron bioavailability from these foods.

DETAILED DESCRIPTION:
Each participant will attend a total of 10 study visits. The first visit will be a screening visit to determine eligibility, and will include the administration of health history and food frequency questionnaires, and a urine pregnancy test. Participant will also be given a ASA24 24-hour dietary recall at visit 1 to return at visit 2. All subsequent visits (2 through 10) will begin with a blood sample (15 mL, or 1 tablespoon, after a 12 hour overnight fast).

Visit 2 will establish the baseline distribution of naturally occurring zinc and iron isotopes in the blood, and will include the administration of water enriched in zinc of a specific naturally-occurring isotopic mass (zinc-68, 4 mg).

Visits 2-5 will be on consecutive days, while Visit 6 will be 14 days following Visit 5. Visits 3 and 4 will include breakfast, lunch, and dinner, each containing a small serving of beans that are enriched in specific isotopic masses of iron and zinc (2 mg each of zinc-67 and iron-57, or 1 mg each of zinc-70 and iron-58). Visits 5 and 6 are for blood sampling, to measure the zinc in blood plasma (Visit 5) and the iron that has reached a 14-day equilibrium in red blood cells (Visit 6). Participants will also be given a ASA24 24-hour dietary recall at visit 6 to return at visit 7.

Visits 6-9 will be on consecutive days, starting 28 days (the approximate length of one menstrual cycle) after Visit 3, while Visit 10 will be 14 days following Visit 9. The 28-day timing is needed to minimize the potential influence of natural variation in circulating hormones, on zinc metabolism. A second urine pregnancy test will be administered on Visit 10, to detect any pregnancies that would have occurred at the time of the study meals 2 weeks prior or earlier. Participants will also be given a ASA24 dietary recall at visit 9 to return at visit 10.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eumenorrheic (regular monthly menstrual cycles of 25-30-days in length)
* BMI 18.5 - 30 kg/m2
* Regular consumer of beans, i.e. ≥ 4 servings per month
* Usual iron intake estimated by Food Frequency Questionnaire to be less than the Recommended Daily Allowance (RDA) of 18 mg/d (8)
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures.

Exclusion Criteria:

* Dislike or allergy to beans
* Self-reported current or recent pregnancy (within the past 12 months)
* Self-reported recent termination of pregnancy (3 months if abortion in 1st or 2nd trimester, or 12 months if in 3rd trimester)
* Self-reported plans to become pregnant during the study period
* Self-reported cancer
* Self-reported surgery without the past 12 months
* Currently taking prescription drugs, other than for contraception, or any nutritional supplements
* Any daily iron supplementation within the past 12 months.
* Currently breastfeeding
* Any medical conditions affecting iron or zinc metabolism (such as hemochromatosis or sickle cell disease)

Ages: 19 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fractional Zinc absorption | 24 hours after first intake
  amount of zinc absorbed and circulating in blood
Fractional Iron absorption | 24 hours after first intake
  amount of iron absorbed and circulating in the blood

SECONDARY OUTCOMES:
Total Zinc absorption | 24 hours after first intake
  total amount of zinc absorbed from meals
Total Iron absorption | 24 hours after first intake
  total amount of iron absorbed from meals

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hall, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No